CLINICAL TRIAL: NCT05064904
Title: Multidiscipline Care for Acute Kidney Injury to Chronic Kidney Disease Transition (Acute Kidney Disease) - a Randomized Controlled Study
Brief Title: Multidiscipline Care for Acute Kidney Disease (AKD)
Acronym: AKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201811079MINC; 201900796A3C502 (Other: Chang Gung Medical Foundation Institutional Review Board)
Record Dates: First submitted 2021-06-11; First posted 2021-10-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Acute Kidney Injury
Keywords: Chronic kidney disease; Acute kidney disease
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The randomization procedure was developed at the WHI Clinical Coordinating Center and implemented locally through a distributed study database, using a randomized permuted block algorithm, stratified by clinical center site, diabetics mellitus and age group.
Who Masked: Participant
Masking Description: The randomization procedure was developed at the WHI Clinical Coordinating Center and implemented locally through a distributed study database, using a randomized permuted block algorithm, stratified by clinical center site, diabetics mellitus and age group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- never received RAAS blockers or multidiscipline consultation before AKI. (Active Comparator): The enrollees assigned to the control group should not receive RAAS blockers or AKD consultation at least in 180 days after index discharge. In addition, these multidiscipline consultation and administration of RAAS blockers are continuing, and results regarding them remain masked. All patients provided written informed consent.
  Interventions: Drug: never received RAAS blockers or received RAAS blockers before AKI.
- had received RAAS blockers and multidiscipline consultation before AKI. (Active Comparator): All enrolled patients are randomly referred to receive comprehensive multidiscipline consultation targeting a glycated hemoglobin level of less than 7.0%, systolic blood-pressure, target, <130 mm Hg, low density lipid (LDL) less than 100mg/dL and control of hyperuricemia less than 7.2mg/deal in male as well as 6.1mg/dl in females. We suggest to adherence to low protein diet achieve the goal of hemoglobin more than 11g/L at 180 day after index discharge.
  Enrollees who are not received renin-angiotensin-aldosterone blockers (RAAS) are randomly assigned to slow kidney function progression by adding RAAS blockers by receiving at least defined daily dose equal to Losartan 50mg or Captopril 25mg bid. The acute kidney disease (AKD) consultation should be transferred at least one time within 90 days after index hospital discharge after withdrawing from dialysis requiring AKI (AKI-D).
  Interventions: Drug: never received RAAS blockers or received RAAS blockers before AKI.

INTERVENTIONS:
Drug: never received RAAS blockers or received RAAS blockers before AKI. — Enrollees who are not received renin-angiotensin-aldosterone blockers (RAAS) are randomly assigned to slow kidney function progression by adding RAAS blockers by receiving at least defined daily dose equal to Losartan 50mg or Captopril 25mg bid. The acute kidney disease (AKD) consultation should be transferred at least one time within 90 days after index hospital discharge after withdrawing from dialysis requiring AKI (AKI-D).
  All enrolled patients are randomly referred to receive comprehensive multidiscipline consultation targeting a glycated hemoglobin level of less than 7.0%, systolic blood-pressure, target, <130 mm Hg, low density lipid (LDL) less than 100mg/dL and control of hyperuricemia less than 7.2mg/deal in male as well as 6.1mg/dl in females. We suggest to adherence to low protein diet achieve the goal of hemoglobin more than 11g/L at 180 day after index discharge.
  Other Names: Multidiscipline consultation

SUMMARY:
The Taiwan Consortium of Acute Kidney Injury and Renal Diseases (TCTC) is leading a clinical trial group in Asia-Pacific to reduce the morbidity and mortality associated with acute kidney injury (AKI). The trial is a double two-by-two factorial design that will collect demographic and clinical information of AKI stage 2, 3, or weaning from dialysis-requiring AKI patients (AKI-D) to explore the epidemiology, risk factors and prognosis of AKI in Taiwan. Patients will be randomized either to add Angiotensin-Converting Enzyme Inhibitors (ACE-I)/Angiotensin II Receptor Blocker (ARB) to slow kidney function progression, or to receive multidisciplinary care. Patients will be followed up for a minimum of 6 months to evaluate kidney function, the predictability of developing chronic kidney disease, end stage renal disease, major cardiovascular events, and mortality.

DETAILED DESCRIPTION:
In the past decade, acute kidney injury (AKI) has emerged as a syndrome of increasing prevalence. Since 2005, hospital-diagnosed cases of AKI have outnumbered those of chronic kidney disease (CKD), and this trend has continued to climb. Patients diagnosed with AKI are at risk for a variety of adverse outcomes, including premature death, morbidity, prolonged hospitalization, and increased medical costs. Potential contributing factors to the development of AKI include pre-existing kidney damage, hemodynamic instability, and the complexity of concurrent medications. As modern medical diagnostic and treatment tools have advanced, the incidence and prevalence of AKI have been steadily rising.

The KDIGO Guideline for AKI recommended that we should diagnose AKI if a given patient has a 6 hour urine amount less than 0.5ml/kg/hr or a serum creatinine elevates more than 0.3mg/dL or 1.5 times greater than baselines. Epidemiology data on hospitalized patients indeed disclosed high risk for adverse events using this classification system and its analogues. However, besides diagnosis, we do not have a useful tool to treat or to help improve patient outcomes Acute kidney injury (AKI) is a common complication that affects nearly 5% of hospitalized patients and 40%-70% of patients in the intensive care unit. AKI requiring dialysis (AKI-D), the most severe type of AKI, is associated with the highest proportion of morbidity and mortality. AKI is associated with a risk of end-stage renal disease (ESRD) that is 13 times as high as the risk among patients without AKI, and the risk of ESRD is 40 times as high if the patients have both AKI and pre-existing chronic kidney disease (CKD). Since AKI is recognized as a risk factor for the development of ESRD, it is crucial to have appropriate protection strategies for the avoidance of further target organ damage and associated mortality in the critical phases of the acute kidney disease (AKD). Patients with Acute Kidney Injury (AKI) requiring dialysis (AKI-D) are associated with the highest proportion of morbidity and mortality. AKI is associated with a thirteen-fold higher risk of end-stage renal disease (ESRD) compared to those without AKI, and a forty-fold higher risk if the patient has both AKI and pre-existing chronic kidney disease (CKD). Given the potential for AKI to lead to ESRD, it is essential to develop strategies to protect the target organs from further damage and associated mortality during the acute phase of AKD. Guyton proposed that the kidneys have a crucial role in determining the chronic level of blood pressure (BP), and studies have validated this hypothesis. Furthermore, hospitalization-associated AKI has been identified as an independent risk factor for the development of elevated BP. Elevated BP is a leading risk factor for global health and cardiovascular disease, making it a key element in the pharmacologic treatment and long-term protection of AKD patients. A retrospective analysis of the ICU database, which included 1551 ICU survivors, 611 of which had AKI during their stay, demonstrated a reduced 1-year mortality in those who had AKI and had been prescribed ACEIs/ARBs.

To address the gap between acute kidney injury (AKI) and chronic kidney disease (CKD), the Kidney Disease: Improving Global Outcomes (KDIGO) AKI Workgroup has proposed the concept of acute kidney disease (AKD). AKD is defined as a glomerular filtration rate (GFR) of less than 60 ml/min/1.73 m2 or evidence of structural kidney damage that has been present for less than 3 months. This concept provides an integrated bridge between AKI and CKD and also emphasizes the concept of partial renal recovery. It may help to raise awareness and create the necessary clinical mechanisms to follow up AKI survivors for the potential progression to CKD, which has been recently highlighted as a missed opportunity for adequate transitions of care. Furthermore, a panel of gut microbiota and biomarkers will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old on the day of index discharge
2. AKI develops during admission, as defined with KDIGO-AKI Guideline, namely, elevation of serum creatinine above 0.3mg/dL within two days, above 1.5 times baseline and ever receives dialysis during this index hospitalization.
3. Patients who has KDIGO-AKI stage 2, 3 or who could wean from dialysis requiring AKI-D in the index hospitalization.

Exclusion Criteria:

1. Baseline estimated glomerular filtration rates (eGFR) less than 5ml/min/1.73m2 or greater than 90ml/min/1.73m2 according to MDRD equation after index discharge.
2. Patients receive further re-dialysis within 90 days after index hospital discharge, who are withdrawal for AKI-D. (sensors)
3. Previous gastrointestinal operations.
4. Patients with major hemorrhage, as defined with acute hemorrhage and requirement of blood transfusion during index admission.
5. Patients with a chronic lung disease requiring non-invasive or invasive positive pressure ventilation.
6. Solid organ or hematological transplantation donors.
7. Evidence of obstructive acute kidney injury.
8. Systolic blood pressure < 110mmHg.
9. Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2024-01-06 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Renal replacement therapy at any time after dialysis | MAKE at 180 days
  Patients will followed up at any time after dialysis.
survival | MAKE at 180 days
  Patients will followed up at any time after death.

SECONDARY OUTCOMES:
Rehospitalization | MAKE at 180 days
  Rehospitalization from myocardial infarction, heart failure, arrhythmia, invasive cardiovascular interventions, cardiovascular causes after noncardiovascular surgery, stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Wu, doctor, Principal Investigator — NTUH
Locations (7):
- Taiwan (7):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Keelung CGMH, Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District